CLINICAL TRIAL: NCT02278107
Title: Evaluation of a Lightweight Nasal Interface and Ventilator for Use by Patients With Respiratory Disease
Brief Title: Evaluation of a Lightweight Nasal Interface and Ventilator in Patients With Respiratory Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: New Aera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: JM-001-2014
Record Dates: First submitted 2014-10-23; First posted 2014-10-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Lung Disease; Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tidal Assist Ventilator System (Experimental): Lightweight, portable, positive pressure ventilator system with proprietary nasal interface. Ventilator is powered by compressed oxygen delivered by cylinder, concentrator, or wall source.
  Interventions: Device: Tidal Assist Ventilator System
- Nasal Cannula Oxygen (Active Comparator): Nasal Cannula Oxygen Standard nasal cannula oxygen at 2-5 liters per minute (LPM) based on patient requirement. Oxygen sources includes cylinder, concentrator, or wall source.
  Interventions: Device: Nasal Cannula Oxygen

INTERVENTIONS:
Device: Tidal Assist Ventilator System — Tidal volume augmentation with supplemental oxygen. Source gas options: cylinder, concentrator, wall.
  Other Names: TAV
  Arms: Tidal Assist Ventilator System
Device: Nasal Cannula Oxygen — Standard oxygen therapy delivered by nasal cannula at 2-5 lpm based on patient requirements. Source gas options: cylinder, concentrator, wall.
  Other Names: Standard oxygen therapy
  Arms: Nasal Cannula Oxygen

SUMMARY:
A preliminary study to evaluate a new nasal interface and portable ventilator system in comparison to standard oxygen therapy in patients with severe chronic lung disease.

DETAILED DESCRIPTION:
An open-label, randomized, controlled, crossover study in patients with severe chronic lung disease to evaluate exercise tolerance compared to standard nasal cannula oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (> 18 years of age) with a diagnosis of severe-to-very severe chronic lung disease
* Participates in a qualified pulmonary rehabilitation program
* Requires constant flow oxygen of ≥ 2 LPM (liters per minute) during exercise
* Able and willing to sign the informed consent
* Ability to be fitted with the test nasal mask and to use the test ventilator system

Exclusion Criteria:

* Requires > 5LPM of constant flow to maintain SpO2> 90% during exercise
* Reports having serious epistaxis within the last 14 days prior to enrollment
* Currently enrolled in another clinical study or has participated within 30 days of enrollment
* Has any condition or abnormality that in the opinion of the Investigators may compromise the participant's safety or the quality of the study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Exercise Endurance Time to Maximum Tolerance | Maximum exercise endurance in minutes, for both treatment arms. Two 4-hr study visits, 1 week apart. Endurance endpoint will be evaluated during a single 4-hr period on Study Visit 2. Each exercise test will be separated by a 1.5 hr rest period.
  Endurance measured on cycle ergometer at predetermined constant work rate. Subjects will exercise to their limit of tolerability (max effort).

SECONDARY OUTCOMES:
Borg 10 Dyspnea Score, Subject reported | Recorded 1-2 min before and every 1 min during exercise testing. Two 4-hr study visits, scheduled 1 week apart. Endpoint will be evaluated during a single 4-hr period on Study Visit 2. Each exercise test will be separated by a 1.5 hr rest period.
  10 point Analog scale
Arterial Oxygen Saturation via Pulse Oximeter (SpO2) | Recorded 1-2 min before and every 1 minute during exercise testing. Two 4-hr study visits, scheduled 1 week apart. Endpoint will be evaluated during a single 4-hr period on Study Visit 2. Each exercise test will be separated by a 1.5 hr rest period.
  SpO2 measured via forehead and finger pulse oximeters
Leg Fatigue, Subject Reported | Recorded 1-2 min before and every 1 min during exercise testing. Two 4-hr study visits, scheduled 1 week apart. Endpoint will be evaluated during a single 4-hr period on Study Visit 2. Each exercise test will be separated by a 1.5 hr rest period.
  10 point Analog scale
Heart Rate | Recorded 1-2 min before and every 1 min during exercise testing. Two 4-hr study visits, scheduled 1 week apart. Endpoint will be evaluated during a single 4-hr period on Study Visit 2. Each exercise test will be separated by a 1.5 hr rest period.
  Heart rate recorded by pulse oximeters
Respiratory Rate | Recorded 1-2 min before and every 1 min during exercise. Evaluated during a single 4-hr period on Study Visit 2. Each exercise test will be separated by a 1.5 hr rest period.
  Respiratory rate recorded by observer
Adverse Events | Two 4-hr study visits, sheduled 1 week apart. Subjects will be monitored for AEs continuously throughuout the study visit. AEs will be monitored and recored during both study visits.
  Monitoring for observed or reported adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kops, MD, Principal Investigator — John Muir Medical Center, Concord Campus

REFERENCES:
- [Background] Porszasz J, Cao R, Morishige R, van Eykern LA, Stenzler A, Casaburi R. Physiologic effects of an ambulatory ventilation system in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2013 Aug 1;188(3):334-42. doi: 10.1164/rccm.201210-1773OC. PMID 23741986
- [Derived] Hilling L, Cayou C, Kops RS, Ameo RA, Morishige RJ, Glezer S, Hill NS. Effect of a Ventilatory Assist Device in Addition to Supplemental Oxygen on Exercise Endurance in Subjects With COPD. Respir Care. 2024 Apr 22;69(5):527-533. doi: 10.4187/respcare.10875. PMID 38199761